CLINICAL TRIAL: NCT03550196
Title: Coronary Artery Bifurcation Revascularization Without kIssing ballOon infLation by rEpoT: The CABRIOLET Study
Brief Title: Coronary Revascularisation by rePOT
Acronym: CABRIOLET
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0877
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Provisional stenting with rePOT technique — All revascularizations have to be performed with complete rePOT technique: initial POT + side branch inflation + final POT. Compliant or semi compliant balloon have to be preferred to inflations. The POT balloon positioning have to be precise as obtain the loose of the parallelism just at the carina cut plan. The rest of the medication or procedure characteristics stay at the discretion of the operator.
  The follow-up will be clinic every years.

SUMMARY:
The presence of a coronary bifurcation complicates percutaneous revascularization. Bifurcation stenting needs to take into account the difference of diameter between proximal and distal vessels and the necessity to limit the side branch obstruction. Provisional stenting techniques with balloon juxtaposition as Kissing Balloon Inflation (KBI) fail to demonstrate a clinical benefits. This is probably explain by the detrimental effect during these technics on the proximal segment with an arterial overstretch. A new sequential technique, named rePOT, demonstrated experimentally a mechanical superiority compared to juxtaposition balloon techniques included KBI. RePOT associates an initial proximal optimizing technique (POT), a side branch inflation and a final POT.

A first clinical study (n=106 patients) confirmed these excellent mechanical results with serial OCT analysis and demonstrated an excellent short term safety. Since 2017, rePOT is recommended in Europe in clinical practice.

This large registry is dedicated to confirm the clinical benefits at long term after bifurcation revascularization with rePOT technique before a large randomise trial.

ELIGIBILITY:
Inclusion Criteria:

* Discovery, during angiography, of a significant coronary lesion (by angiographic or functional assessment) including a bifurcation under a provisional stenting strategy. Bifurcation have to be significant according to the operator and the coronary anatomy (but the side branch diameter have to be greater than 1.75mm)
* Stable lesion without high thrombus burden
* Patient agreement to study participation and ≥ 18 years

Exclusion Criteria:

* Complex lesion or anatomy requiring revascularization strategy with more than one stent
* Contraindication to a double platelet anti-aggregation ≥ 6mois (recommended implantation of active stent)
* Unstable patient according to the operator (used of hemodynamic drug support, mechanical ventilation)
* Indication of cardiac surgery.
* Lesion culprit in ST- or non ST-elevation myocardial infarction <12h.
* High thrombus burden in angiography or endocoronary imaging (IVUS, OCT).
* Pregnancy, loose of legal right
* Other interventional study participation <30 jours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient with stable coronary lesion interesting a bifurcation with indication of revascularization (angiographique or functional) by provisional stenting technique can be included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Long-term clinical benefits after revascularization of coronary bifurcations by the technique of provisional stenting rePOT. | At 12 months
  Number of deaths
Long-term clinical benefits after revascularization of coronary bifurcations by the technique of provisional stenting rePOT. | At 12 months
  Number of myocardial infections
Long-term clinical benefits after revascularization of coronary bifurcations by the technique of provisional stenting rePOT. | At 12 months
  Number of stent thrombosis
Long-term clinical benefits after revascularization of coronary bifurcations by the technique of provisional stenting rePOT. | At 12 months
  Number of target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Département de cardiologie Clinique Axium, Aix-en-Provence
  - Fédération de cardiologie médicale - Hôpital Cardiologique Louis Pradel - Hospices civils de Lyon, Bron
  - Département de cardiologie Hôpital Gabriel Montpied CHU de Clermont Ferrand, Clermont-Ferrand
  - Département de cardiologie CHU de Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No